CLINICAL TRIAL: NCT05623761
Title: The Effect of Toothpastes Based on Alkaline Thermal Water With and Without Fluorinated Derivative on Gingivitis, Dentin Hypersensitivity, and Oral Hygiene: a Randomized Clinical Trial
Brief Title: Toothpastes With Thermal Water for Oral Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18081212
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Gingivitis; Dentin Hypersensitivity
Keywords: gingivitis; dentin sensitivity; thermal water; toothpaste; fluoride
MeSH Terms: conditions — Gingivitis; Dentin Sensitivity | interventions — Fluorides

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, two-arm parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation concealment will be performed using sealed containers numbered by a "third party" (person who will not participate in the study). The toothpastes in white bottles without any titles will be placed in the containers. Each patient will receive a sealed container with a toothpaste on enrolment. Neither patients nor researchers will be aware of the type of the toothpaste used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - toothpaste containing thermal water of Castera-Verduzan and 1450 ppm Sodium fluoride (Active Comparator): Subjects will receive thermal water/sodium fluoride toothpaste (BUCCOTHERM® Sensitive Gums with Fluoride)
  Interventions: Drug: BUCCOTHERM® Sensitive Gums with Fluoride
- Group 2 - toothpaste containing thermal water of Castera-Verduzan (Active Comparator): Subjects will receive thermal water toothpaste (BUCCOTHERM® Sensitive Gums Fluoride-Free)
  Interventions: Drug: BUCCOTHERM® Sensitive Gums Fluoride-Free

INTERVENTIONS:
Drug: BUCCOTHERM® Sensitive Gums with Fluoride — Toothbrushing using standardised technique and pear-sized amount of toothpaste BUCCOTHERM® Sensitive Gums with Fluoride twice daily for 1 month.
  Arms: Group 1 - toothpaste containing thermal water of Castera-Verduzan and 1450 ppm Sodium fluoride
Drug: BUCCOTHERM® Sensitive Gums Fluoride-Free — Toothbrushing using standardised technique and pear-sized amount of toothpaste BUCCOTHERM® Sensitive Gums Fluoride-Free twice daily for 1 month.
  Arms: Group 2 - toothpaste containing thermal water of Castera-Verduzan

SUMMARY:
The aim of the study is to compare the effect of toothpastes containing thermal water of Castera-Verduzan with 1450 ppm fluoride and without fluorinated derivatives on oral hygiene, gingivitis, and dentin hypersensitivity in young adults.

DETAILED DESCRIPTION:
This will be a double-blind, randomized, two-arm parallel-group study of the effect of toothpastes containing thermal water of Castera-Verduzan with 1450 ppm fluoride and without fluorinated derivatives. The groups will include adults with gingivitis and dentinal hypersensitivity (DH) diagnosed clinically. To assess the effect of the toothpastes, the following parameters will be used: gingival health (modified gingival index, MGI; gingival bleeding index, BI), dentin sensitivity (Shiff's index, VAS), oral hygiene level (Navi-Rustogi index), and salivary pH.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20-25 years
* signed an approved Informed Consent Form, authorizing the participation in the trial and the use of the results of the trial for educational purposes and for the publication
* the diagnosis of gingivitis stated clinically
* at least one tooth with the diagnosis of dentin hypersensitivity stated clinically

Exclusion Criteria:

* medical and pharmacotherapeutic histories that may compromise the protocol (pregnancy or breastfeeding, psychiatric disorders, allergies to toothpastes ingredients, eating disorders)
* systemic conditions that are etiologic to dentin hypersensitivity (e.g., chronic acid regurgitation)

history of chemotherapy or radiotherapy

* taking antibiotic, anti-inflammatory, or anti-coagulant medications 4 weeks prior to or after the baseline visit
* oral mucosa pathology
* periodontal surgery in the preceding 3 months
* orthodontic appliance treatment within previous 3 months
* teeth or supporting structures with any other painful pathology or defects
* taking any other agents for DH management 4 weeks prior to or after the baseline visit
* extensively restored teeth and those with restorations extending into the

cervical area

* dental bleaching within previous 3 months
* subject withdrawal of consent
* subject is not compliant with study procedures
* adverse Event that in the opinion of the Investigator would be in the best interest

of the subject to discontinue study participation

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of gingival inflammation by Modified Gingival Index (MGI) | 4 weeks after the baseline
  MGI is used to assess visual symptoms of gingivitis on facial and lingual surfaces of each scorable tooth (whole mouth). Two scores are recorded buccally/labially, two scores lingually/palatally. Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-4). Scoring is performed using standard dental light:0=absence of inflammation,1=mild inflammation;slight change in color,little change in color; little change in texture of any portion of the marginal or papillary gingival unit,2=mild inflammation; criteria as above plus the entire marginal or papillar gingival unit,3=moderate inflammation;glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit,4=severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit,spontaneous bleeding,congestion,or ulceration. Lower scores indicate better results.
Evaluation of gingival inflammation by Bleeding Inde | 4 weeks after the baseline
  BI is used to assess bleeding elicited on probing as a measure of gingival condition. Gingivae are air dried and examiner assesses bleeding using a probe which is gently inserted into gingival crevice to depth of app 1 mm and run around tooth (angle of app 60 deg to long axis of tooth), gently stretching epithelium while sweeping from interproximal to interproximal along sulcular epithelium. BI is assessed on facial and lingual gingival surfaces of each scorable tooth (whole mouth). 3 scores are recorded buccally/ labially, 3scores lingually/ palatally. All scorable teeth in one quadrant are probed first (app 30 sec) before recording number of gingival units which bleed. Values are presented as means across all tooth surfaces with minimum and maximum scores in agreement with minimum and maximum index values (i.e., 0-2). BI score:0=no bleeding after 30 sec, 1=bleeding upon probing after 30 sec,2=immediate bleeding. Lower scores indicate better results.
Evaluation of DH according to Shiff sensitivity score | 4 weeks after the baseline
  First, the tooth is isolated by the cotton roll from the adjacent teeth. Next, a blast of air from a standard dental unit syringe at 60 ± 5 psi at 18-22 °C is directed onto the exposed middle 1/3 buccal surface for 1 s at a distance of approximately 10 mm. Then, each patient reports the sensitivity he/she sensed using Schiff Cold Air Sensitivity scale scored from 0 to 3: score "0" means no response, score "1" means response without request of discontinuation of stimulus, score "2" means response with request of discontinuation of stimulus, and score "3" means pain with request of discontinuation of stimuli. Lower scores indicate better results.

SECONDARY OUTCOMES:
Evaluation of oral hygiene level according to Navi-Rustogi index | 4 weeks after the baseline
  Nine sites per facial and lingual tooth surface are assessed, for a maximum 504 sites total (excluding 3rd molars, crowns, and surfaces with cervical restorations). Disclosed plaque is scored in each tooth area as follows: 0 = Absent; and 1 = Present. A mean plaque index (MPI) is calculated for each subject on a whole mouth basis. Lower scores indicate better results.
Evaluation of salivary pH | 3 minutes after baseline (after toothbrushing)
  Unstimulated 5 ml whole saliva sample is collected in morning from 10 am to 11 am, two hours after the last meal. Participants refrain from eating, drinking, smoking, or conducting oral hygiene procedures for a minimum of 90 min prior to salivary collection. Participants are comfortably seated, are asked to avoid swallowing saliva and asked to lean forward and spit all the saliva they produced into a graduated test tube until the required volume is collected. The pH is determined immediately after the collection using a digital pH-meter.

CONTACTS AND LOCATIONS:
Overall Officials: Irina M Makeeva, Principal Investigator — +79037280722
Locations (1):
- Institute of Dentistry of Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makeeva IM, Polyakova MA, Doroshina VY, Turkina AY, Babina KS, Arakelyan MG. [Comparative effectiveness of therapeutic toothpastes with fluoride and hydroxyapatite]. Stomatologiia (Mosk). 2018;97(5):34-40. doi: 10.17116/stomat20189705134. Russian. PMID 30346419
- [Background] Makeeva IM, Polyakova MA, Doroshina VY, Sokhova IA, Arakelyan MG, Makeeva MK. [Efficiency of paste and suspension with nano-hydroxyapatite on the sensitivity of teeth with gingival recession]. Stomatologiia (Mosk). 2018;97(4):23-27. doi: 10.17116/stomat20189704123. Russian. PMID 30199063
- [Background] Polyakova M, Sokhova I, Doroshina V, Arakelyan M, Novozhilova N, Babina K. The Effect of Toothpastes Containing Hydroxyapatite, Fluoroapatite, and Zn-Mg-hydroxyapatite Nanocrystals on Dentin Hypersensitivity: A Randomized Clinical Trial. J Int Soc Prev Community Dent. 2022 Apr 8;12(2):252-259. doi: 10.4103/jispcd.JISPCD_333_21. eCollection 2022 Mar-Apr. PMID 35462739